CLINICAL TRIAL: NCT04148534
Title: Intraoperative Monitoring of Facial Nerve in Patients Undergoing Cerbellopontine Angle Tumer Resection Using Partial Versus no Neuromuscular Block
Brief Title: Compare the Operating Condition of Two Levels of Muscle Relaxation on Facial Nerve MEP Monitoring in CPA Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Magdy Gaber (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Muhammad Magdy Gaber, Ass lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: D-4-2019
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cerebellopontine Angle Tumor
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- muscle relaxant (Active Comparator): patient who will receive muscle relaxant, patients will receive rocronium infusion by (5 mcg/kg/min) , maintain partial NMB TOF count 2 and targeting BIS = (40-60)
  Interventions: Drug: Rocroniom, Non Depolarizing Muscle Relaxant
- without muscle relaxant (Placebo Comparator): patient who will not receive muscle relaxant, will recieve normal saline targeting BIS = 40-60.
  Interventions: Drug: Rocroniom, Non Depolarizing Muscle Relaxant

INTERVENTIONS:
Drug: Rocroniom, Non Depolarizing Muscle Relaxant — compare the operating condition of two different levels of muscle relaxation on facial nerve monitoring using transcranial motor evocked potential in CPA surgery
  Other Names: Nerve stimulator for train of four assessment; BIS bispectral index

SUMMARY:
compare the operating condition of two different levels of muscle relaxation on facial nerve monitoring using transcranial motor evocked potential in CPA surgery .

* To Estimate End to start facial nerve MEP amplitude ratio
* To determine the effect of neuromuscular relaxant degrees on recovery and
* Assessment of propofol doses needed for enhancement of early recovery and ambulation.

DETAILED DESCRIPTION:
40 Patients aged from 18-60 years old undergoing Cerebellopontine angle surgery. Patients will be one of two groups: Both Induction will be accomplished with fentanyl, propofol , rocronium infusion will be given randomly to one of the groups.

Depth of anaesthesia, neurotransmitter monitoring and facial nerve neurophysiological monitoring will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between >18 and<60.
* Patients scheduled for neurosurgical CPA surgeries
* Ability to sign the consent
* ASA classification I, II

Exclusion Criteria:

* ASA > II
* Hemodynamically unstable
* Disease affecting neuromuscular transmission (myasthenia gravies ...etc.)
* GCS < 15.
* Any cardiac patient (ischemic heart disease - cardiomyopathy...etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
End to start facial nerve MEP amplitude ratio. | 6 to 8 month
  TCMEP recording will begin (1) prior to skin incision as baseline amplitude before muscle relaxant be taken for intubation (2) at Dural closure and end \start amplitude ratio will be calculated.

SECONDARY OUTCOMES:
number of hypotension episodes and the use of vasopressors | 6 to 8 month
  hemodynamic condition
Total volume of propofol and fentanyl infused | 6 to 8 month
  Calculate dose consumption

CONTACTS AND LOCATIONS:
Overall Officials: Cairo university, Principal Investigator — Cairo university faculty of medicine research ethical committee
Locations (1):
- Cairo university medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No